CLINICAL TRIAL: NCT01879319
Title: A Multicenter, Randomized Study in Subjects With Primary Hypercholesterolemia or Mixed Dyslipidemia to Assess Subjects' Ability to Administer a Full Dose of Evolocumab (AMG 145) in Home-use, Using Either a 3.5 mL Personal Injector or a Prefilled Autoinjector/Pen.
Brief Title: Study to Assess in Home Use of Evolocumab (AMG 145) Administration Using Either an Automated Mini-doser or a Prefilled Autoinjector/Pen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120356
Record Dates: First submitted 2013-06-13; First posted 2013-06-17 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Primary Hypercholesterolemia; Mixed Dyslipidemia
Keywords: LDL-C, triglycerides, high cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evolocumab AMD (Experimental): Participants received evolocumab 420 mg once a month subcutaneously using an automated mini-doser (AMD) (one 3.5 mL injection) for 8 weeks (Day 1, Week 4, and Week 8). Participants self-administered evolocumab in the clinic on Day 1 under supervision and then self-administered in a home setting at Weeks 4 and 8.
  Interventions: Biological: Evolocumab AMD
- Evolocumab AI/pen (Experimental): Participants received evolocumab 420 mg once a month subcutaneously using an autoinjector/pen (AI/pen) (three 1.0 mL injections) for 8 weeks (Day 1, Week 4, and Week 8). Participants self-administered evolocumab in the clinic on Day 1 under supervision and then self-administered in a home setting at Weeks 4 and 8.
  Interventions: Biological: Evolocumab AI/pen

INTERVENTIONS:
Biological: Evolocumab AMD — Evolocumab subcutaneous injection using a single use, disposable AMD containing 3.5 mL deliverable volume.
  Other Names: AMG 145; Repatha
  Arms: Evolocumab AMD
Biological: Evolocumab AI/pen — Evolocumab subcutaneous injection using a handheld mechanical (spring-based) prefilled AI/Pen, each containing 1.0 mL deliverable volume.
  Other Names: AMG-145; Repatha
  Arms: Evolocumab AI/pen

SUMMARY:
The primary objective of this study was to assess users' ability to administer a full dose of evolocumab in a home-use setting using either an automated mini-doser (AMD) or autoinjector/pen (AI/pen).

ELIGIBILITY:
Inclusion Criteria:

* Fasting LDL-C at screening > 85 mg/dL
* Fasting triglycerides less than or equal to 400 mg/dL (4.5 mmol/L)

Exclusion Criteria:

* New York Heart Association (NYHA) III or IV heart failure
* Uncontrolled cardiac arrhythmia
* Uncontrolled hypertension
* Type 1 diabetes or poorly controlled type 2 diabetes
* Uncontrolled hypothyroidism or hyperthyroidism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2013-07-11 (Actual); Primary Completion 2013-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (26):
- United States (21):
  - Research Site, Phoenix, Arizona
  - Research Site, Encino, California
  - Research Site, Thousand Oaks, California
  - Research Site, Tustin, California
  - Research Site, Ventura, California
  - Research Site, Port Charlotte, Florida
  - Research Site, Saint Augustine, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Lexington, Kentucky
  - Research Site, Lewiston, Maine
  - Research Site, Ayer, Massachusetts
  - Research Site, Manlius, New York
  - Research Site, Cadiz, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Lansdale, Pennsylvania
  - Research Site, Jackson, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
- Canada (5):
  - Research Site, Burnaby, British Columbia
  - Research Site, London, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Pointe-Claire, Quebec

REFERENCES:
- [Background] Boccara F, Dent R, Ruilope L, Valensi P. Practical Considerations for the Use of Subcutaneous Treatment in the Management of Dyslipidaemia. Adv Ther. 2017 Aug;34(8):1876-1896. doi: 10.1007/s12325-017-0586-8. Epub 2017 Jul 17. PMID 28717862
- [Background] Kasichayanula S, Grover A, Emery MG, Gibbs MA, Somaratne R, Wasserman SM, Gibbs JP. Clinical Pharmacokinetics and Pharmacodynamics of Evolocumab, a PCSK9 Inhibitor. Clin Pharmacokinet. 2018 Jul;57(7):769-779. doi: 10.1007/s40262-017-0620-7. PMID 29353350
- [Background] Toth PP, Descamps O, Genest J, Sattar N, Preiss D, Dent R, Djedjos C, Wu Y, Geller M, Uhart M, Somaratne R, Wasserman SM; PROFICIO Investigators. Pooled Safety Analysis of Evolocumab in Over 6000 Patients From Double-Blind and Open-Label Extension Studies. Circulation. 2017 May 9;135(19):1819-1831. doi: 10.1161/CIRCULATIONAHA.116.025233. Epub 2017 Mar 1. PMID 28249876
- [Background] Toth PP, Jones SR, Monsalvo ML, Elliott-Davey M, Lopez JAG, Banach M. Effect of Evolocumab on Non-High-Density Lipoprotein Cholesterol, Apolipoprotein B, and Lipoprotein(a): A Pooled Analysis of Phase 2 and Phase 3 Studies. J Am Heart Assoc. 2020 Mar 3;9(5):e014129. doi: 10.1161/JAHA.119.014129. Epub 2020 Mar 2. PMID 32114889
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were men and women ≥ 18 and ≤ 80 years of age with fasting low-density lipoprotein cholesterol (LDL-C) ≥ 85 mg/dL, fasting triglycerides ≤ 400 mg/dL and on a stable dose of a statin with or without ezetimibe for at least 4 weeks. The first patient enrolled on 11 July 2013 and the last patient enrolled on 20 September 2013.
Pre-assignment Details: Randomization was stratified on the basis of screening LDL-C concentration (< 130 mg/dL [3.4 mmol/L] or ≥ 130 mg/dL). Participants were trained by study site staff to prepare and self-administer the study drug.
Period: Overall Study
Arm/Group | Evolocumab AMD | Evolocumab AI/Pen
Started | 82 | 82
Received Treatment | 82 | 82
Completed | 80 | 77
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 5

BASELINE CHARACTERISTICS:
Population: Full analysis set (all randomized participants who received at least 1 dose of study drug).
Groups:
- Evolocumab AMD: Participants received evolocumab 420 mg once a month subcutaneously using an automated mini-doser (AMD) (one 3.5 mL injection) for 8 weeks (Day 1, Week 4, and Week 8).
- Evolocumab AI/Pen: Participants received evolocumab 420 mg once a month subcutaneously using an autoinjector/pen (AI/pen) (three 1.0 mL injections) for 8 weeks (Day 1, Week 4, and Week 8).
- Total: Total of all reporting groups
Arm/Group | Evolocumab AMD | Evolocumab AI/Pen | Total
Number analyzed (Participants) | 82 | 82 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (10.5) | 59.2 (10.0) | 59.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 39 | 78
  Male | 43 | 43 | 86
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 4 | 3 | 7
  Black or African American | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 69 | 75 | 144
  Other | 2 | 0 | 2
  Mixed Race | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 78 | 76 | 154
Stratification Factor: LDL-C Level [Number; unit: participants]
  < 130 mg/dL | 60 | 59 | 119
  ≥ 130 mg/dL | 22 | 23 | 45
LDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] | 115.3 (27.0) | 117.3 (23.9) | 116.3 (25.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Full Administration of Evolocumab at Both Weeks 4 and 8
Description: Self-administration of evolocumab was assessed by a telephone interview at Weeks 4 and 8. Each participant was asked about all attempted injection(s) and if the injection was administered in part, full, or none at all. Results only include full administrations that occurred inside the prespecified visit window.
Time Frame: Weeks 4 and 8
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Evolocumab AMD | Evolocumab AI/Pen
Number analyzed (Participants) | 82 | 82
Percentage of participants | 93.9 [86.5 to 97.4] | 91.5 [83.4 to 95.8]
Statistical Analysis 1: Comparison: Evolocumab AMD vs Evolocumab AI/Pen; Test type: Superiority or Other; Treatment Difference = -2.4, 95% CI 2-sided [-11.2 to 6.1]

2. Secondary Outcome: Percent Change From Baseline in LDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Evolocumab AMD | Evolocumab AI/Pen
Number analyzed (Participants) | 82 | 82
percent change | -67.9 (2.4) | -64.5 (2.4)
Statistical Analysis 1: Comparison: Evolocumab AMD vs Evolocumab AI/Pen; Test type: Superiority or Other; LS Mean Treatment Difference = 3.4, 95% CI 2-sided [-2.9 to 9.7], Standard Error of Mean 3.2

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 28 days after last study drug administration (up to 12 weeks)
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Evolocumab AMD | Evolocumab AI/Pen
Serious Adverse Events (participants affected / at risk) | 0/82 | 1/82
Other Adverse Events (participants affected / at risk) | 0/82 | 0/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Evolocumab AMD (N=82) | Evolocumab AI/Pen (N=82)
Deep vein thrombosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.